CLINICAL TRIAL: NCT04105218
Title: The Effect of Exercise on Sleep Quality and Nocturnal Fat Oxidation in Individuals With Metabolic Syndrome
Brief Title: Exercise, Sleep Quality and Nocturnal Fat Oxidation in Metabolic Syndrome
Acronym: ExerciZzz
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Personnel resources required to conduct study are no longer available. Study was terminated due to lack of resources
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18-0369
Record Dates: First submitted 2019-09-03; First posted 2019-09-26 (Actual); Results first posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Metabolic Syndrome; PreDiabetes; Hypertension; Obesity; Hyperlipidemias
MeSH Terms: conditions — Metabolic Syndrome; Prediabetic State; Hypertension; Obesity; Hyperlipidemias | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evening Exercise (Experimental): Participants will arrive in the Clinical and Translation Research Center (CTRC) and enter the whole room calorimeter approximately 1 hour after arrival. During the evening exercise condition, participants will perform 45-minutes of moderate intensity continuous exercise on a treadmill 12 hours after habitual wake time in the evening. Participants will begin with a warm-up for 5 minutes at 2.0-2.5 mph. Heart rate will be monitored continuously with a heart rate monitor. Participants will maintain heart rate at 65% of age-predicted maximum heart rate. Throughout the day, participants will be required to eat the standardized meals provided at breakfast lunch and dinner. At the time of bed, participants will be instructed to turn off the lights, lay down in bed and to refrain from using electronic devices. In the morning, a metabolic test will be performed and melatonin levels will be measured in the saliva
  Interventions: Behavioral: Exercise
- Control (Placebo Comparator): Participants will arrive in the Clinical and Translation Research Center (CTRC) in the morning within 2 hours of their habitual wake time. Participants will enter the whole room calorimeter approximately 1 hour after arriving at the CTRC. Throughout the day, participants will be required to eat the standardized meals provided at breakfast lunch and dinner. At the time of bed, participants will be instructed to turn off the lights, lay down in bed and to refrain from using electronic devices. In the morning, a metabolic test will be performed and melatonin levels will be measured in the saliva
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants will perform 4 study visits over 1-3 months. The 1st study visit is a screening visit, during which eligibility will be determined. During the 2nd visit, resting metabolic rate (RMR) and body composition will be measured. Participants will also perform a submaximal exercise test. Prior to each condition, habitual sleep/wake patterns will then be measured for 1 week. Participants will then perform each of the 2 study conditions (evening exercise and control) in randomized order with at least a 1-week washout period between conditions. Females will be studied during the luteal phase to control for potential confounding effects of hormonal variations across the menstrual cycle.

SUMMARY:
The purpose of the Exerci-Zzz Study is to learn more about how the time of day that exercise is performed influences sleep quality and fat metabolism overnight in adults with metabolic syndrome. In this study, exercise will be performed in the early evening and the investigators will measure participants' sleep quality and fat metabolism overnight in a metabolic room. The total study will take approximately 2-3 months to complete.

Enrolled participants will complete 2 study conditions (evening exercise and control) in a metabolic room. Each of these visits will last 30 hours and require that the participant stay in the metabolic room. During the evening exercise participants will be asked to perform exercise in the early evening. Finally, during the control condition participants will be asked spend the day in the metabolic room (no exercise performed during this condition). During each of these conditions, the investigators will measure participant sleep quality and fat metabolism overnight. In the morning, the investigators will perform a metabolic test to assess the responses of certain hormones. Findings from this study will identify how exercise influences novel contributors to metabolic syndrome (sleep quality and nocturnal metabolism) and shed light on some potential mechanisms to explain the variability in exercise responses.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS) is a major risk factor for many chronic diseases, including diabetes and cardiovascular disease. Sleep is recognized a risk factor for many of the conditions comprising MetS (e.g. high blood sugars, obesity). Interestingly, fat metabolism during your sleep is important for regulating several key components of health, like risk of obesity and glucose tolerance. While exercise is recognized as a health enhancing behavior to reduce the risk of many chronic diseases, the effect of exercise on sleep quality and nocturnal fat metabolism is largely unknown. This study plans to learn more about how the time of day that you perform exercise influences sleep quality and fat metabolism overnight in adults with metabolic syndrome. In this study, exercise will be performed in the early evening and the investigators will measure your sleep quality and fat metabolism overnight in our metabolic room. Findings from this study will identify how exercise influences novel contributors to metabolic syndrome (sleep quality and nocturnal metabolism) and shed light on some potential mechanisms to explain the variability in exercise responses.

ELIGIBILITY:
Inclusion Criteria:

* not currently meeting physical activity guidelines (<150 minutes moderate to vigorous physical activity per week);
* weight stable (<5% change in weight over the last 6 months);
* habitual sleep duration of 7-8 hours and consistent sleep/wake schedule (<1 hour variation night-to-night).

Exclusion Criteria:

* body mass index >35.0 kg/m2; pregnancy;
* post-menopausal status in women, confirmed by absences of menses for >1 year and elevated follicular stimulating hormone concentrations (>50 mIU/mL); women on oral contraceptives;
* self-reported diabetes, cardiovascular disease, or sleep disorder;
* untreated hyper/hypothyroidism, cancer;
* inability to perform moderate to vigorous treadmill exercise;
* shiftwork

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Blankenship, PhD, Principal Investigator — jennifer.blankenship@cuanschutz.edu
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
We currently do not have a plan to share IDP

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study screened 91 individuals and enrolled 12 participants, however, due to the multiple COVID-19 clinical research shutdowns, only one of the participants was able to complete any of the inpatient study visits (though she withdrew after this visit). During the COVID19 shutdowns, 6 of the 12 participants withdrew from the study primarily due to increased childcare responsibilities. 3 participants failed screening tests during the baseline visit.
Groups:
- Evening Exercise Condition --> Control Condition: Participants will arrive in the Clinical and Translation Research Center (CTRC) and enter the whole room calorimeter approximately 1 hour after arrival. Participants will perform 45-min of moderate intensity continuous exercise on a treadmill 12 hours after habitual wake time in the evening. Participants will begin with a warm-up for 5 minutes at 2.0-2.5 mph. Heart rate will be monitored continuously with a heart rate monitor. Participants will maintain heart rate at 65% of age-predicted maximum heart rate. Throughout the day, participants will be required to eat the standardized meals provided at breakfast lunch and dinner. At the time of bed, participants will be instructed to turn off the lights, lay down in bed and to refrain from using electronic devices. In the morning, a metabolic test will be performed and melatonin levels will be measured in the saliva
  Exercise: Participants will perform 4 study visits over 1-3 months. The 1st study visit is a screening visit, during which eligibility will be determined. During the 2nd visit, resting metabolic rate (RMR) and body composition will be measured. Participants will also perform a submaximal exercise test. Prior to each condition, habitual sleep/wake patterns will then be measured for 1 week. Participants will then perform each of the 2 study conditions (evening exercise and control) in randomized order with at least a 1-week washout period between conditions. Females will be studied during the luteal phase to control
- Control Condition --> Evening Exercise Condition: Participants will arrive in the Clinical and Translation Research Center (CTRC) in the morning within 2 hours of their habitual wake time. Participants will enter the whole room calorimeter approximately 1 hour after arriving at the CTRC. Throughout the day, participants will be required to eat the standardized meals provided at breakfast lunch and dinner. At the time of bed, participants will be instructed to turn off the lights, lay down in bed and to refrain from using electronic devices. In the morning, a metabolic test will be performed and melatonin levels will be measured in the saliva
  Exercise: Participants will perform 4 study visits over 1-3 months. The 1st study visit is a screening visit, during which eligibility will be determined. During the 2nd visit, resting metabolic rate (RMR) and body composition will be measured. Participants will also perform a submaximal exercise test. Prior to each condition, habitual sleep/wake patterns will then be measured for 1 week. Participants will then perform each of the 2 study conditions (evening exercise and control) in randomized order with at least a 1-week washout period between conditions. Females will be studied during the luteal phase to control for potential confounding effects of hormonal variations across the menstrual cycle.
Period: Overall Study
Arm/Group | Evening Exercise Condition --> Control Condition | Control Condition --> Evening Exercise Condition
Started | 6 | 6
Completed First Condition | 0 | 1
Completed Second Condition | 0 | 0
Completed | 0 | 0
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Study was terminated; unable to complete study visits | 1 | 3
Not completed — Failed screening tests | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Evening Exercise Condition --> Control Condition | Control Condition --> Evening Exercise Condition | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 12
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (6.2) | 31.67 (5.8) | 33 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Nocturnal FFA Concentrations
Description: Free Fatty Acids (FFA) concentrations
Time Frame: 8-hours
Population: Study terminated before sufficient outcome measure data could be collected to make analysis possible for this outcome measure. No data was able to be analyzed.
Groups:
- Evening Exercise: Participants will arrive in the Clinical and Translation Research Center (CTRC) and enter the whole room calorimeter approximately 1 hour after arrival. Participants will perform 45-min of moderate intensity continuous exercise on a treadmill 12 hours after habitual wake time in the evening. Participants will begin with a warm-up for 5 minutes at 2.0-2.5 mph. Heart rate will be monitored continuously with a heart rate monitor. Participants will maintain heart rate at 65% of age-predicted maximum heart rate. Throughout the day, participants will be required to eat the standardized meals provided at breakfast lunch and dinner. At the time of bed, participants will be instructed to turn off the lights, lay down in bed and to refrain from using electronic devices. In the morning, a metabolic test will be performed and melatonin levels will be measured in the saliva
  Exercise: Participants will perform 4 study visits over 1-3 months. The 1st study visit is a screening visit, during which eligibility will be determined. During the 2nd visit, resting metabolic rate (RMR) and body composition will be measured. Participants will also perform a submaximal exercise test. Prior to each condition, habitual sleep/wake patterns will then be measured for 1 week. Participants will then perform each of the 2 study conditions (evening exercise and control) in randomized order with at least a 1-week washout period between conditions. Females will be studied during the luteal phase to control
Arm/Group | Evening Exercise | Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Nocturnal Fat Oxidation
Description: Total fat oxidation (measured by whole room calorimeter)
Time Frame: 8-hours
Population: as for outcome 1
Arm/Group | Evening Exercise | Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Nocturnal Glucose and Insulin Concentrations
Description: Nocturnal glycemic control
Time Frame: 8-hours
Population: as for outcome 1
Arm/Group | Evening Exercise | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Sleep Quality (Percent Time in Slow Wave Sleep [SWS])
Description: Time spent in slow wave sleep
Time Frame: 8-hours
Population: as for outcome 1
Arm/Group | Evening Exercise | Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Sleep Latency
Description: Time spent to fall asleep
Time Frame: 8-hours
Population: as for outcome 1
Arm/Group | Evening Exercise | Control
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Sleep Interruptions
Description: Wake after sleep onset [WASO]
Time Frame: 8-hours
Population: as for outcome 1
Arm/Group | Evening Exercise | Control
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Dietary Fat Oxidation
Description: Measured using a palmitate stable isotope tracer at breakfast
Time Frame: 24-hours
Population: as for outcome 1
Arm/Group | Evening Exercise | Control
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Distal/Proximal Temperature Gradient
Description: Skin temperature at distal and proximal body locations
Time Frame: 24-hours
Population: as for outcome 1
Arm/Group | Evening Exercise | Control
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Melatonin Offset
Description: Melatonin concentrations
Time Frame: First 5 hours of waking (after study condition)
Population: as for outcome 1
Arm/Group | Evening Exercise | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to12 months
Description: Adverse event definition is the same as clinicaltrials.gov
Arm/Group | Evening Exercise | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT04105218/Prot_SAP_000.pdf